CLINICAL TRIAL: NCT05683977
Title: EvaluatioN of durvALumab Utilization and Effectiveness for First Line Extensive Stage Small Cell Lung Cancer. Prospective Cohort of Extensive Stage Small Cell Lung Cancer Patients Treated With Durvalumab Associated With Platinum-etoposide Chemotherapy
Brief Title: A French Real-life Study: EvaluatioN of durvALumab Utilization and Effectiveness for First Line Extensive Stage Small Cell Lung Cancer.
Acronym: ARSENAL
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Kappa Santé (Industry)
Responsible Party: Sponsor
Other Study IDs: D419QR00014
Record Dates: First submitted 2022-10-26; First posted 2023-01-13 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — durvalumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: durvalumab — Visits will be completed at W0 (durvalumab in combination with chemotherapy initiation) and at regular visits approximately every 6 weeks during the induction period (durvalumab + PE) (W6 and W12), then every two months during the maintenance period (durvalumab alone) for the first year and every three months up to the end of follow-up or the final visit at M36.

SUMMARY:
Small cell lung cancer (SCLC), characterized by rapid proliferation, high growth fraction and early development of metastases, is the most aggressive form of lung cancer. In 2021, an estimated 2.3 million people around the world are diagnosed with lung cancer. In France, in 2018, with 46 363 new cases and 33 117 deaths, lung cancer represented the second most common cancer and the first cause of death from cancer. Among those, SCLC represented 10,8% of all new lung diagnosis, and about two thirds presented at the extensive stage (ES-SCLC).

Since last three decades, standard treatment in ES-SCLC is based on combination chemotherapy with a platinum agent and etoposide in first-line with or without concurrent radiation therapy. Then, the second-line of treatment is topotecan, with few results in terms of response rates and survival rate. However, the emergence of immune checkpoint inhibitors targeting the programmed cell death receptor-1 (PD-1)/PD-ligand 1 (PD-L1) pathway, having an important role in immune regulation became an alternative method in the management and care of disease. Indeed, recent studies have shown an overall survival (OS) benefit for patients with ES-SCLC treated in first line with a combination of platinum-etoposide and immune checkpoint inhibitors. Atezolizumab (Tecentriq®, Roche) and durvalumab (Imfinzi®, AstraZeneca), two anti-Programmed death-ligand 1 (PD-L1) antibodies, delivered positive phase III results, respectively through the Impower-133 and CASPIAN studies, and were granted European market authorisations.

Durvalumab is approved for use in combination with etoposide and either carboplatin or cisplatin for the first-line treatment of patients with ES-SCLC. On March 10, 2020 French health authorities allowed durvalumab utilization in this setting through a national "early access program" (Autorisation Temporaire d'Utilisation "de cohorte" - ATUc), thus preceding the European market authorization (August 28, 2020). Since 2020 October 1st, durvalumab is used as a post ATU treatment. Since 2020, French AURA treatment guidelines for SCLC have referenced durvalumab in combination with chemotherapy as a first-line treatment option for patients with ES-SCLC.

Whereas the safety and efficacy of the durvalumab have been evaluated in a clinical trial, data are required to further evaluate the use of durvalumab in real-life condition and in less selected population than in clinical trials.

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC), characterized by rapid proliferation, high growth fraction and early development of metastases, is the most aggressive form of lung cancer. SCLC is a relatively rare but really aggressive tumour accounting for 10-15% of all newly diagnosed lung cancer. In 2021, an estimated 2.3 million people around the world are diagnosed with lung cancer . In France, in 2018, with 46 363 new cases and 33 117 deaths, lung cancer represented the second most common cancer and the first cause of death from cancer. Among those, SCLC represented 10,8% of all new lung diagnosis, and about two thirds presented at the extensive stage (ES-SCLC).

Between 2010 and 2018, the incidence rate increased of 0,3 % per year in men. In contrast, from 1990 to 2018, the incidence increased more dramatically among women, with an increase of 5% in average per year. The 5-year survival rate for all people with all types of lung cancer is 21%. The 5-year survival rate is 17% and 24% for men and women, respectively. For SCLC, due to the rapid proliferation and high growth fraction associated to early development of metastases in the disease course (most commonly to the brain, liver, or bone), the 5-year survival rate is low at 10%. Therefore, SCLC is the most lethal lung cancer subtype. Most cases of SCLC develop in patients aged 60-80 years and the estimated overall death rate is 25,000-30,000 per year in United States. More than 90% of patients with SCLC are elderly and have heavy smoking histories.

SCLC is defined histologically as "a malignant epithelial tumour consisting of small cells with scant cytoplasm, ill-defined cell borders, finely granular nuclear chromatin, and absent or inconspicuous nucleoli", assessed by imaging techniques such as computerized tomography (CT), positron emission tomography (PET) and magnetic resonance imaging (MRI).

The Veterans' Administration Lung Study Group (VALG) staging system is usually used in the clinic routine to stage SCLC. Two categories represent SCLC, limited stage (LS) and extensive stage (ES). Limited-stage small-cell lung cancer (LS-SCLC) is defined as tumour confined to one hemithorax, with or without regional lymph-node involvement, which can be safely encompassed in a tolerable radiation field, corresponding at stage I to III of TNM system. ES-SCLC is defined as disease that cannot be safely encompassed in a tolerable radiation field, corresponding to stage IV of TNM system.

The management of SCLC is complicated by aggressiveness and substantial comorbidities, and impaired performance status. According to ESMO guidelines (2021), as well as in the French guidelines from Auvergne Rhone Alpes region, the standard management design of SCLC is described and outlined in Figure 1.

Since last three decades, standard treatment in ES-SCLC is based on combination chemotherapy with a platinum agent and etoposide in first-line with or without concurrent radiation therapy. Then, the second-line of treatment is topotecan, with few results in term of response rates and survival rate.

However, the emergence of immune checkpoint inhibitors targeting the programmed cell death receptor-1 (PD-1)/PD-ligand 1 (PD-L1) pathway, having an important role in immune regulation became an alternative method in the management and care of disease. Indeed, recent studies have shown an overall survival (OS) benefit for patients with ES-SCLC treated in first line with a combination of platinum-etoposide and immune checkpoint inhibitors. Atezolizumab (Tecentriq®, Roche) and durvalumab (Imfinzi®, AstraZeneca), two anti-Programmed death-ligand 1 (PD-L1) antibodies, delivered positive phase III results, respectively through the Impower-133 and CASPIAN studies, and were granted European market authorisations.

Durvalumab (Imfinzi®, AstraZeneca), a fully human monoclonal antibody against programmed cell death-ligand 1 (PD-L1), is approved for use in combination with etoposide and either carboplatin or cisplatin for the first-line treatment of patients with ES-SCLC. On March 10, 2020 French health authorities allowed durvalumab utilization in this setting through a national "early access program" (Autorisation Temporaire d'Utilisation "de cohorte" - ATUc), thus preceding the European market authorization (August 28, 2020). Since 2020 October 1st, durvalumab is used as a post ATU treatment.

Since 2020, French AURA treatment guidelines for SCLC have referenced durvalumab in combination with chemotherapy as one of the first-line treatment options for patients with ES-SCLC based on evidence from the CASPIAN phase III international randomized clinical trial, which demonstrated that adding durvalumab to chemotherapy significantly improved the median overall survival (mOS; hazard ratio: 0.73, 95% confidence interval (CI): 0.59-0.91) over chemotherapy alone.

Results from this CASPIAN study was recently updated with an assessment of 3-year overall survival. As of 2021 March, with a median follow-up 39.4 months, durvalumab plus chemotherapy continued to demonstrate a significant improvement OS versus chemotherapy alone (P = 0.0003). Authors concluded three times more patients were estimated to be alive at 3 years when treated with durvalumab plus chemotherapy versus chemotherapy, with the majority still receiving durvalumab at data cut-off, further establishing durvalumab plus chemotherapy as first-line standard of care for ES-SCLC.

To date, durvalumab has thus been available to first-line ES-SCLC patients and clinicians have the choice between atezolizumab + carboplatin-etoposide, durvalumab + carbo- or cisplatin-etoposide, and carbo- or cisplatin-etoposide alone.

Whereas the safety and efficacy of the durvalumab have been evaluated in clinical trial, data are required to further evaluate the use of durvalumab in real-life condition and in less selected population than in clinical trials, while it received EMA approval in 2020. Some studies with durvalumab were performed in real-life, but only for non-SCLC.

This observational uncontrolled prospective cohort study is conducted to complement evidence from the CASPIAN clinical trial and generate real-world evidence. There is indeed a need to describe durvalumab use in the clinical practice for the treatment of first-line ES-SCLC patients and broaden the CASPIAN results to real-life setting in France.

Therefore, the aim of this study is to describe of platinum-etoposide and durvalumab real-life utilization and effectiveness for first line ES-SCLC.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (at least 18 years of age at time of treatment decision),
* Patients with histologically or cytologically proven SCLC and extensive disease according to the Veterans Administration Lung Study Group (VALSG) classification or TNM staging (Brierley et al, 2017) before durvalumab + platinum-etoposide treatment*,
* Patients newly treated in first line with durvalumab + platinum-etoposide**,
* Patients informed and not opposed to participating in the study.

Exclusion Criteria:

* Patients with contraindications to receiving durvalumab + platinum-etoposide,
* Patients participating in another interventional clinical trial for first line ES-SCLC.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Total population: all patients enrolled
  * Safety analysis set: the safety population will be defined as all patients who receive at least one infusion of durvalumab.
  * Full analysis set: the full analysis set will comprise all patients who receive at least one infusion of durvalumab and meet eligibility criteria.
  * Follow up analysis set: it will comprise all patients of the full analysis set who have at least one follow up visit completed.
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
The time to first line treatment discontinuation (TTD). | TTD is defined as the time from the index date to the date of last durvalumab infusion (+3 weeks during induction period and +4 weeks during maintenance period) or date of death (up to 36 months)).
  For patients who start durvalumab at a later cycle than first cycle PE, the index date will be the first infusion of PE.
  If the treatment is stopped during the first phase of 4 to 6 cycles (induction) with a new re- start of durvalumab and PE, the treatment will be considered as temporary stop. If the treatment is stopped during the durvalumab maintenance with a re-start of durvalumab in monotherapy, the treatment will be also considered as temporary stop.
  Durvalumab will be considered definitely discontinued when the maintenance phase with durvalumab in monotherapy is stopped and results in a new administration of PE (+/-durvalumab) (subsequent treatment line).
  For patients still receiving durvalumab at the end of follow-up or when they are lost to follow-up, TTD will be right-censored at the last recorded day of ongoing durvalumab treatment.

SECONDARY OUTCOMES:
Real-world Overall Survival (rwOS) | rwOS rate at 1, 2 and 3 years (rwOS1y, rwOS2y, rwOS3y)
  rwOS is defined as the time from index date (date of first infusion of durvalumab and/ or platinum-etoposide) to date of death due to any cause. rwOS will be censored on the last date patient is known to be alive.
  rwOS rate at 1, 2 and 3 years (rwOS1y, rwOS2y, rwOS3y) and median real-world overall survival (mrwOS) will be assessed.
Real world Progression Free Survival (rwPFS) | rwPFS rate at 6, 12, 18, 24 and 36 months (rwPFS6m, rwPFS12m, rwPF18m, rwPFS24m, rwPFS36m) up to 36 months.
  rwPFS is defined as the time from index date (date of first infusion of durvalumab and/ or platinum-etoposide) to the date of disease progression as assessed by physicians or the date of death, whichever occurs first. rwPFS will be censored on the date of last follow-up.
  The rwPFS date will be based on the investigator's judgement. The real-world progression may be based on radiological evaluation or clinical judgement, or other measure to compensate absence of RECIST criteria.
  rwPFS rate at 6, 12, 18, 24 and 36 months (rwPFS6m, rwPFS12m, rwPF18m, rwPFS24m, rwPFS36m) and median rwPFS (mrwPFS) will be assessed.
Patient individual best response | From the start of treatment until disease progression (up to 36 months)..
  The tumour response will be assessed by investigator as Complete response (CR), Partial response (PR), Stable disease (SD), Progressive disease (PD). The patient individual best response is defined as the best response recorded from the start of treatment until disease progression.
  The proportion of patients with a CR as best response, with a PR as best response, with SD as best response and with PD as best response will be assessed.
Overall response rate (ORR) | From the start of treatment until disease progression (up to 36 months).
  ORR is defined as proportion of patients with at least one complete response (CR) or partial response (PR) at least one visit (Paz Ares et al, 2019).
Disease control rate (DCR) | At the end of follow-up (up to 36 months)
  DCR is defined as the proportion of patients with at least one complete response (CR), partial response (PR) or stable disease.
Time to second real-world progression (rwPFS2) | rwPFS2 (up to 36 months)
  rwPFS2 is defined as the time from index date (date of first infusion of durvalumab and/ or platinum-etoposide) to the second record of disease progression determined by physicians' assessment, or death. rwPFS2 will be right-censored at the date of last follow-up.
Sociodemographics characteristics at durvalumab + platinum-etoposide initiation | At baseline
  Age
Describe patient history prior to durvalumab initiation | Before durvalumab initiation
  Proportion of patients with previous history of cancer, Proportion of patients with history of paraneoplastic syndromes, Proportion of patients with history of auto-immune disease (including past, stabilized or active disease, disease duration), Proportion of patient treated with antibiotics, corticosteroids or other immunosuppressive therapy in the last 4 weeks before treatment initiation.
  Treatment history at durvalumab + platinum-etoposide initiation will be described in terms of:
  Proportion of patients with previous SCLC anti-cancer therapy (for limited and extensive stage),
  Proportion of patients with previous auto-immune disease associated treatment, Proportion of patients with previous non cancer therapies of interest (immunosuppressive therapy, nephrotoxic and anti-inflammatory drugs, antibiotherapy, corticosteroid therapy, supportive treatments).
Describe the safety profile of durvalumab + chemotherapy (PE) (treatment-related AE). | At the end of follow-up (up to 36 months).
  Safety profile of durvalumab + platinum-etoposide will be described in terms of:
  * Incidence rate of grade ≥3 durvalumab -related according to Common Terminology Criteria for Adverse Events (CTCAE),
  * Incidence rate of durvalumab -related immune-related AEs (imAE),
  * Incidence rate of SAEs, AESIs, AEs resulting in treatment modification,
  * Incidence rate of AEs resulting in treatment discontinuation,
Sociodemographics characteristics at durvalumab + platinum-etoposide initiation | At baseline
  Gender
Sociodemographics characteristics at durvalumab + platinum-etoposide initiation | At baseline
  BMI
Sociodemographics characteristics at durvalumab + platinum-etoposide initiation | At baseline
  Smoking status
Clinical characteristics at durvalumab + platinum-etoposide initiation | At baseline
  * Duration between initial SCLC diagnosis and ES-SCLC for patients with first diagnosis at limited stage,
  * Duration between initial ES-SCLC diagnosis and treatment initiation,
Clinical characteristics at durvalumab + platinum-etoposide initiation | At baseline
  - Disease stage at tumour diagnosis (limited or extensive stage; number of metastatic sites) and at baseline,
Clinical characteristics at durvalumab + platinum-etoposide initiation | At baseline
  - Actual number and localization of metastases at baseline including brain metastases (symptomatic or asymptomatic, treated or not), bone metastases (extension), and liver metastases,
Clinical characteristics at durvalumab + platinum-etoposide initiation | At baseline
  - Performance status at baseline (before durvalumab initiation),
Clinical characteristics at durvalumab + platinum-etoposide initiation | At baseline
  Comorbidities.
Describe patient history prior to durvalumab initiation | Before durvalumab discontinuation
  Time from discontinuation of the last treatment received for limited stage to start of first treatment for extensive stage
Safety profile of durvalumab + chemotherapy (PE) (treatment-related AE). | At the end of follow-up (up to 36 months).
  - Description of concomitant treatments including nephrotoxic and steroids-immunosuppressive drugs used to manage durvalumab related adverse events.

OTHER OUTCOMES:
Describe the nature and explore the impact of different sequential therapeutical strategies on patient outcomes. | At the end of follow-up (up to 36 months)
  The impact of different sequential therapeutical strategies (including local and systemic treatments) on patient outcomes will be described in terms of:
  - Treatment pathways description (sequences description, duration of sequences),
Explore disease characteristics, that may influence the progression of cancer and/or response to durvalumab + platinum etoposide treatment | At the end of follow-up (up to 36 months).
  The association between clinical and biomolecular disease characteristics and cancer progression or response to treatment will be investigated.
Time between chemotherapy and durvalumab initiation: | Between chemotherapy and durvalumab initiation (up to 1 year)
  Time between chemotherapy and durvalumab initiation is defined as the time from date of first infusion of platinum etoposide to the date of first infusion of durvalumab.
Dosing regimen and scheme | At the end of follow-up (up to 36 months)
  * Proportion of patients receiving durvalumab-etoposide-cisplatin,
  * . Proportion of patients receiving durvalumab-etoposide-carboplatin,
  * Proportion of patients receiving the combination durvalumab plus PE at first infusion (first cycle),
  * Proportion of patients receiving PE at first infusion and durvalumab at a later cycle (if later, initiation cycle),
Chemotherapy cycles description | At the end of follow-up (up to 36 months)
  * Proportion of patients treated with 4 cycles/ 6 cycles before maintenance period,
  * Proportion of patients with doses modifications during treatment, description of the changes,
  * Proportion of patients with delayed cycles and reason for delay.
Number of durvalumab cycles | At the end of follow-up -up to 36 months)
  * Number of cycles with durvalumab in combination with PE (induction period),
  * Number of cycles with durvalumab in monotherapy (maintenance period),
Duration of treatment | At the end of follow-up (up to 36 months).
  Mean and median duration of first line treatment from the date of first infusion of durvalumab and /or PE to the date of last infusion of durvalumab.
Time to first subsequent therapy (TFST) | At the end of the follow-up (up to 36 months).
  TFST is defined as the time from the index date (date of first infusion of durvalumab and/ or platinum-etoposide) to the date of subsequent therapy or the date of death. For patients still receiving durvalumab at the end of follow-up, TFST will be right-censored at the last recorded day of ongoing durvalumab treatment.
Time to second subsequent therapy (TSST) | At the end of follow-up (up to 36 months).
  TSST is defined as the time from the index date (date of first infusion of durvalumab and/ or platinum-etoposide) to the date of second subsequent therapy or date of death. For patients still receiving durvalumab at the end of follow-up, TSST will be right-censored at the last recorded day of ongoing durvalumab treatment.
Local and supportive treatments | At the end of follow-up (up to 36 months).
  * Proportion of patients with mediastinal irradiation while on durvalumab treatment,
  * Proportion of patients with prophylactic cranial irradiation while on durvalumab treatment,
  * Proportion of patients with other irradiation while on durvalumab treatment,
  * Proportion of patients with surgery while on durvalumab treatment,
  * Proportion of patients with GCS-F while on durvalumab treatment,
  * Proportion of patients with EPO while on durvalumab treatment,
  * Proportion of patients with phosphonate while on durvalumab treatment,
Describe the nature and explore the impact of different sequential therapeutical strategies on patient outcomes. | At the end of follow-up (up to 36 months)
  - Pattern of tumor progression, rwPFS2, TFST, TSST).
Describe the nature and explore the impact of different sequential therapeutical strategies on patient outcomes. | At the end of follow-up (up to 36 months)
  - Treatment effectiveness (ORR, DCR, mrwOS, mrwPFS, mrwPFS2, TFST, TSST).
Dosing regimen and scheme | At the end of follow-up (up to 36 months)
  * Description of dosage for durvalumab plus PE at initiation
  * Description of reasons for platinum salt choice (better tolerance, better efficacy, hospital protocol, patient status, age, other),
Number of chemotherapy cycles | At the end of follow-up (up to 36 months)
  Number of cycles with platinum-etoposide,
Chemotherapy cycles delays | At the end of follow-up (up to 36 months)
  - Time between each cycle,
Durvalumab cycles delays | At the end of follow-up (up to 36 months)
  - Time between each cycle,
Description of durvalumab cycles | At the end of follow-up (up to 36 months)
  - Proportion of patients with delayed cycles and reason for delay.
Local and supportive treatments timeline | At the end of follow-up (up to 36 months)
  Time between the end of induction period and the first local treatment (mediastinal irradiation or prophylactic cranial irradiation).

CONTACTS AND LOCATIONS:
Locations (31):
- France (31):
  - Research Site, Angers
  - Research Site, Argenteuil
  - Research Site, Avignon
  - Research Site, Bayonne
  - Research Site, Bordeaux
  - Research Site, Clermont-Ferrand
  - Research Site, Créteil
  - Research Site, Dijon
  - Research Site, Epagny Metz-Tessy
  - Research Site, Évreux
  - Research Site, Gleizé
  - Research Site, La Roche-sur-Yon
  - Research Site, La Rochelle
  - Research Site, Le Chesnay-Rocquencourt
  - Research Site, Limoges
  - Research Site, Marseille
  - Research Site, Nancy
  - Research Site, Nîmes
  - Research Site, Osny
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Saint-Etienne
  - Research Site, Saint-Grégoire
  - Research Site, Saint-Quentin
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Valenciennes
  - Research Site, Vannes
  - Research Site, Villeurbanne

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Avrillon V, Daniel C, Boisselier P, Le Pechoux C, Chouaid C. Nationwide Real-Life Safety and Treatment Exposure Data on Durvalumab After Concurrent Chemoradiotherapy in Unresectable Stage III, Locally Advanced, Non-small Cell Lung Cancer: Analysis of Patients Enrolled in the French Early Access Program. Lung. 2022 Feb;200(1):95-105. doi: 10.1007/s00408-022-00511-8. Epub 2022 Feb 9. PMID 35141799
- [Background] Carter BW, Glisson BS, Truong MT, Erasmus JJ. Small cell lung carcinoma: staging, imaging, and treatment considerations. Radiographics. 2014 Oct;34(6):1707-21. doi: 10.1148/rg.346140178. PMID 25310425
- [Background] Eberhardt WE, Mitchell A, Crowley J, Kondo H, Kim YT, Turrisi A 3rd, Goldstraw P, Rami-Porta R; International Association for Study of Lung Cancer Staging and Prognostic Factors Committee, Advisory Board Members, and Participating Institutions. The IASLC Lung Cancer Staging Project: Proposals for the Revision of the M Descriptors in the Forthcoming Eighth Edition of the TNM Classification of Lung Cancer. J Thorac Oncol. 2015 Nov;10(11):1515-22. doi: 10.1097/JTO.0000000000000673. PMID 26536193
- [Background] Evans WK, Shepherd FA, Feld R, Osoba D, Dang P, Deboer G. VP-16 and cisplatin as first-line therapy for small-cell lung cancer. J Clin Oncol. 1985 Nov;3(11):1471-7. doi: 10.1200/JCO.1985.3.11.1471. PMID 2997406
- [Background] Goldstraw P, Chansky K, Crowley J, Rami-Porta R, Asamura H, Eberhardt WE, Nicholson AG, Groome P, Mitchell A, Bolejack V; International Association for the Study of Lung Cancer Staging and Prognostic Factors Committee, Advisory Boards, and Participating Institutions; International Association for the Study of Lung Cancer Staging and Prognostic Factors Committee Advisory Boards and Participating Institutions. The IASLC Lung Cancer Staging Project: Proposals for Revision of the TNM Stage Groupings in the Forthcoming (Eighth) Edition of the TNM Classification for Lung Cancer. J Thorac Oncol. 2016 Jan;11(1):39-51. doi: 10.1016/j.jtho.2015.09.009. PMID 26762738
- [Background] Horn L, Mansfield AS, Szczesna A, Havel L, Krzakowski M, Hochmair MJ, Huemer F, Losonczy G, Johnson ML, Nishio M, Reck M, Mok T, Lam S, Shames DS, Liu J, Ding B, Lopez-Chavez A, Kabbinavar F, Lin W, Sandler A, Liu SV; IMpower133 Study Group. First-Line Atezolizumab plus Chemotherapy in Extensive-Stage Small-Cell Lung Cancer. N Engl J Med. 2018 Dec 6;379(23):2220-2229. doi: 10.1056/NEJMoa1809064. Epub 2018 Sep 25. PMID 30280641
- [Background] Nicholson AG, Chansky K, Crowley J, Beyruti R, Kubota K, Turrisi A, Eberhardt WE, van Meerbeeck J, Rami-Porta R; Staging and Prognostic Factors Committee, Advisory Boards, and Participating Institutions; Staging and Prognostic Factors Committee Advisory Boards and Participating Institutions. The International Association for the Study of Lung Cancer Lung Cancer Staging Project: Proposals for the Revision of the Clinical and Pathologic Staging of Small Cell Lung Cancer in the Forthcoming Eighth Edition of the TNM Classification for Lung Cancer. J Thorac Oncol. 2016 Mar;11(3):300-11. doi: 10.1016/j.jtho.2015.10.008. Epub 2015 Dec 24. PMID 26723244
- [Background] Paz-Ares L, Chen Y, Reinmuth N, Hotta K, Trukhin D, Statsenko G, Hochmair MJ, Ozguroglu M, Ji JH, Garassino MC, Voitko O, Poltoratskiy A, Musso E, Havel L, Bondarenko I, Losonczy G, Conev N, Mann H, Dalvi TB, Jiang H, Goldman JW. Durvalumab, with or without tremelimumab, plus platinum-etoposide in first-line treatment of extensive-stage small-cell lung cancer: 3-year overall survival update from CASPIAN. ESMO Open. 2022 Apr;7(2):100408. doi: 10.1016/j.esmoop.2022.100408. Epub 2022 Mar 10. PMID 35279527
- [Background] Paz-Ares L, Dvorkin M, Chen Y, Reinmuth N, Hotta K, Trukhin D, Statsenko G, Hochmair MJ, Ozguroglu M, Ji JH, Voitko O, Poltoratskiy A, Ponce S, Verderame F, Havel L, Bondarenko I, Kazarnowicz A, Losonczy G, Conev NV, Armstrong J, Byrne N, Shire N, Jiang H, Goldman JW; CASPIAN investigators. Durvalumab plus platinum-etoposide versus platinum-etoposide in first-line treatment of extensive-stage small-cell lung cancer (CASPIAN): a randomised, controlled, open-label, phase 3 trial. Lancet. 2019 Nov 23;394(10212):1929-1939. doi: 10.1016/S0140-6736(19)32222-6. Epub 2019 Oct 4. PMID 31590988
- [Background] Travis WD, Asamura H, Bankier AA, Beasley MB, Detterbeck F, Flieder DB, Goo JM, MacMahon H, Naidich D, Nicholson AG, Powell CA, Prokop M, Rami-Porta R, Rusch V, van Schil P, Yatabe Y; International Association for the Study of Lung Cancer Staging and Prognostic Factors Committee and Advisory Board Members. The IASLC Lung Cancer Staging Project: Proposals for Coding T Categories for Subsolid Nodules and Assessment of Tumor Size in Part-Solid Tumors in the Forthcoming Eighth Edition of the TNM Classification of Lung Cancer. J Thorac Oncol. 2016 Aug;11(8):1204-1223. doi: 10.1016/j.jtho.2016.03.025. Epub 2016 Apr 21. PMID 27107787
- [Background] Wang S, Zimmermann S, Parikh K, Mansfield AS, Adjei AA. Current Diagnosis and Management of Small-Cell Lung Cancer. Mayo Clin Proc. 2019 Aug;94(8):1599-1622. doi: 10.1016/j.mayocp.2019.01.034. PMID 31378235
- [Background] Wang S, Tang J, Sun T, Zheng X, Li J, Sun H, Zhou X, Zhou C, Zhang H, Cheng Z, Ma H, Sun H. Survival changes in patients with small cell lung cancer and disparities between different sexes, socioeconomic statuses and ages. Sci Rep. 2017 May 2;7(1):1339. doi: 10.1038/s41598-017-01571-0. PMID 28465554
- [Background] Falchero L, Tissot C, Duruisseaux M, Souquet P-J,Planchard D , et le comité de rédaction des référentiels Auvergne Rhône-Alpes en oncologie thoracique. Référentiel Cancer Bronchique à petites Cellules : actualisation 2022. ARISTOT 2022.
- [Background] APM News. L'activité de prise en charge des cancers dans les établissements Français en 2018 (Infographie). 21/11/2019.
- [Background] Brierley JD, Gospodarowicz MK, Wittekind C, et al, eds. TNM Classification of Malignant Tumours. 8th ed. Oxford, UK: Wiley Blackwell; 2017.
- [Background] Deffossez, G. Estimations nationales de l'incidence et de la mortalité par cancer en France métropolitaine entre 1990 et 2018. Volume 1 - Tumeurs solides. 2019.
- [Background] Navada S, Lai P, Schwartz AG, and Kalemkerian GP (2006). Temporal trends in small cell lung cancer: Analysis of the national Surveillance, Epidemiology, and End Results database (abstract 7082). J Clin Oncol 24(18_suppl), 7082-7082.
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Oronsky B, Reid TR, Oronsky A, Carter CA. What's New in SCLC? A Review. Neoplasia. 2017 Oct;19(10):842-847. doi: 10.1016/j.neo.2017.07.007. Epub 2017 Sep 6. PMID 28888101
- [Result] Armeni P, Borsoi L, Fornaro G, Jommi C, Grossi F, Costa F. Cost-effectiveness and Net Monetary Benefit of Durvalumab Consolidation Therapy Versus No Consolidation Therapy After Chemoradiotherapy in Stage III Non-small Cell Lung Cancer in the Italian National Health Service. Clin Ther. 2020 May;42(5):830-847. doi: 10.1016/j.clinthera.2020.03.012. Epub 2020 Apr 27. PMID 32354495
- See also: Dewolf, M. et al. Référentiel sur le cancer bronchique à petites cellules - Actualisation 2021. ONCOLOGIK.2021. Accessible to: http://oncologik.fr/referentiels/rrc/cancer-bronchique-a-petites-cellules (13.07.21) (2021). — http://oncologik.fr/referentiels/rrc/cancer-bronchique-a-petites-cellules
- See also: ASCO 2021 — https://www.cancer.net/cancer-types/lung-cancer-non-small-cell/statistics.